CLINICAL TRIAL: NCT03777137
Title: Investigation of the Effect of Transcranial Magnetic Stimulation of Several Sites in the Brain Upon Experimental Pain
Brief Title: The Effect of Transcutaneous Magnetic Stimulation on Acute Pain.
Status: Withdrawn | Type: Observational
Why Stopped: Expired in the IRB
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00084600
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Pain Perception
Keywords: Brain network for pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMS during heat pain stimuli: This is a single institution, single-blinded, long-term exploratory study using participant as his/her own control to evaluate and compare the analgesic effect of experimental heat pain of TMS during early versus late times on a vigilance behaviors toward pain (CPT, Continuous Performance Task). Vigilance behaviors include errors, reaction times and activation.
  Interventions: Behavioral: TMS (Rapid2, Magstim Corp)

INTERVENTIONS:
Behavioral: TMS (Rapid2, Magstim Corp) — Volunteers will take a telephone screening questionnaire and those meeting inclusion criteria will attend their first visit. Those signing the consent will have a T1 weighted MRI scan to localize sites in the brain to be stimulated with TMS. The subjects will then have four visits at intervals of two weeks; each visit will have a TMS intervention including SITE1, SITE2, SITE3, and SITE4. The sequence of the testing TMS four different visits (SITE1 to SITE4) will be randomly assigned among stimulation sites Medial Frontal (MF), Dorsal Lateral Frontal (DL), Primary motor cortex (M1) and Interparietal Sulcus (Sham) and counterbalanced across subjects (see Diagram below). During each of visits 2 to 5, each participant will undergo baseline Quantitative Sensory Testing (QST), followed by a TMS intervention, and then by repeat QST. QST will consist of pain thresholds for contact heat.

SUMMARY:
This is a single institution, single-blinded, long-term exploratory study using participant as his/her own control to evaluate and compare the potential analgesic effect on experimental heat pain of Transcutaneous Magnetic Stimulation (TMS). TMS will be delivered by a commercially available device (Rapid2, Magstim Corp) at three different cortical target sites and one sham target site in healthy participants 18-88 years of age. The quantitative evaluation measure is the change in the painful heat threshold Quantitative Sensory Testing (QST) of thresholds for cutaneous heat stimuli before and after TMS.

DETAILED DESCRIPTION:
After subjects contact the office to express interest in being involved with this protocol, subjects will take the telephone screening questionnaire. Those who meet inclusion criteria with no exclusions will come for first visit. At this visit, subjects will discuss and sign the consent form, and have a one sequence MRI scan which is used to localize sites in the brain to be stimulated with TMS.

The subjects will then have four visits at intervals of two weeks; each visit will have TMS intervention designated (SITE1), (SITE2), (SITE3), and (SITE4). TMS will be applied each of four sites (SITE1, SITE2, SITE3, and SITE4) which will be randomly assigned among stimulation sites Medial Frontal (MF), Dorsolateral Frontal (DL), Primary Motor Cortex (M1 and superior Interparietal sulcus (Sham) and counterbalanced across subjects (see Diagram below).

During each of visits 2 to 5, the participant will undergo baseline Quantitative Sensory Testing (QST), followed by TMS stimulation and then by repeat QST. QST will consist of pain thresholds for cutaneous hot stimuli. Visits 2 through 5 will last for approximately 1 hour each and will occur at two-week intervals. The total study duration will be 50 days for each subject. Study enrollment will last for three years and total study duration will be four years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman 18-80 years of age;
* Possess the ability to understand study procedures and comply with them for the entire length of the study;
* Women of childbearing age must use contraception for duration of study.

Exclusion Criteria:

* History of diagnosis of heart disease, increased intracranial pressure, or structural abnormalities of the brain (e.g. tumor);
* History of epilepsy, seizure disorder, neurologic disease, cranial trauma or head surgery, or implanted hardware (including cardiac pacemakers, cardiac lines, medication pumps, or stimulators);
* Family history of seizures;
* Presence of metal anywhere deep to or on the skull (excluding the mouth);
* Any current or recent (<6 weeks) or planned (within duration of study period) use of any of the following medications: imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, ketamine, gamma-hydroxybutyrate (GHB), and theophylline;
* History of peripheral neuropathy, e.g. Diabetic Neuropathy;
* Women who are pregnant or women of childbearing capacity who may become pregnant (i.e. not using contraception);
* Volunteers with communication disorders or non-English speakers;
* Current drug or alcohol use or dependence that, in the opinion of the investigators, would interfere with adherence to study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will include healthy men and women between 18 and 80 years of age with no history or family history of seizures. In addition, subjects cannot be taking pro-epileptic medications or have metal objects in the head except the mouth, as described in the telephone screening questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Contact Heat Pain Temperature Threshold Change | Entire duration of study, approximately five years
  The contact heat thermal thermode will be used to measure heat pain thresholds (in degrees centigrade) before and after each stimulation site.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Lenz, Principal Investigator — Department of Neurosurgery, JHU
Locations (1):
- Hopkiins Functional Neurosurgery Lab, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This data may be shared with other investigators in Baltimore studying pain perception by techniques including brain imaging or psychophysics.

REFERENCES:
- [Background] . Lenz FA, Casey KL, Jones EG, Willis WD, The human pain system: experimental and clinical perspectives. Cambridge, UK ; New York: Cambridge University Press; 2010.